CLINICAL TRIAL: NCT01665274
Title: A Randomized Single Center Controlled Study of Perioperative Chemotherapy of Oxaliplatin Combined With Capecitabine (XELOX) Versus XELOX as Post-operative Chemotherapy in Advanced Gastric Adenocarcinoma With D2 Dissection
Brief Title: Efficiency of XELOX Neoadjuvant Chemotherapy in Gastric Cancer
Acronym: repeat
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: we are working on a larger similar multicenter cinical trials as a participant.so in order to avoid conflicts of interest, we have to suspended this project.
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yingwei Xue, Chief of Gastrointestinal Surgery, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCPCT1205/repeat
Record Dates: First submitted 2012-08-05; First posted 2012-08-15 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Gastric Cancer
Keywords: xelox; advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XELOX adjuvant group (Active Comparator): D2 resection
  XELOX (Drug: Capecitabine 1,000 mg/m² twice daily. Film coated tablets of 500 mg. d1-14 q3w Drug: Oxaliplatin IV infusion, 130mg/m² d1 q3w) 6 cycles
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Procedure: D2 resection
- XELOX neoadjuvant (Experimental): XELOX (Drug: Capecitabine 1,000 mg/m² twice daily. Film coated tablets of 500 mg. d1-14 q3w Drug: Oxaliplatin IV infusion, 130mg/m² d1 q3w) 3 cycles chemotherapy before operation.
  D2 resection
  After operation:
  CR/PR: XELOX (Drug: Capecitabine 1,000 mg/m² twice daily. Film coated tablets of 500 mg. d1-14 q3w Drug: Oxaliplatin IV infusion, 130mg/m² d1 q3w) 3 cycles chemotherapy after operation. SD/PD:,ST(Drug: S-1，40-75mg twice daily. d1-14 q3w Drug: Paclitaxel IV infusion 135mg/m2 d1; q3w) 3 cycles chemotherapy after operation.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Procedure: D2 resection

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1,000 mg/m² twice daily, d1-14, q3w
  Other Names: xeloda
Drug: Oxaliplatin — Oxaliplatin IV infusion, 130mg/m² d1, q3w
  Other Names: eloxatin
Procedure: D2 resection — D2 resection

SUMMARY:
The purpose of this study is to demonstrate that capecitabine/oxaliplatin as perioperative chemotherapy is superior or not to operation directly for locally advanced gastric cancer in terms of 3 year disease-free survival (DFS) rate.

DETAILED DESCRIPTION:
The patients of gastric cancer have been divided into two parts in random.The test group receive perioperative chemotherapy (XELOX) six cycles and the control group administrate the same program after operation. The two groups have the same staging and eligibility criteria.The 3 year disease-free survival (DFS) rate and 5 year overall survival (OS) rate maybe the last evaluation standard.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status of ≥60 %.
* Histologically confirmed gastric adenocarcinoma, staged pathologically or clinically, stage cT2-4N+M0, and cT4N0M0.
* Patients had to have adequate renal function (serum creatinine ≤1 times the upper limit of normal [ULN]), hepatic function (total bilirubin ≤1·5 times the ULN, aspartate or alanine aminotransferase ≤2·5 times the ULN, alkaline phosphatase ≤2·5 times the ULN, Serum albumin ≥30g/L), and haematological function (absolute neutrophil count ≥1·5×10⁹/L and platelet count ≥100×10⁹/L)

Exclusion Criteria:

* Pregnant or lactating women.
* According to the AJCC TMN 7.0, Any evidence of metastatic (TxNxM1) patients(including presence of tumor cells in the ascites).
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy except corticosteroids, for the currently treated gastric cancer.
* Has uncontrolled epilepsy, central nervous system diseases or mental disorders of history.
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, New York Heart Association (NYHA) grade II or greater congestive heart failure or serious cardiac arrhythmia requiring medication or myocardial infarction within the last 12 months.
* Lack of physical integrity of the upper gastrointestinal tract or those who have malabsorption syndrome likely to influence absorption of capecitabine, or inability to take oral medication.
* Known peripheral neuropathy ≥ CTCAEv3 grade 1 (Common Terminology for Adverse Events). Absence of deep tendon reflexes as the sole neurologic abnormality does not render the patient ineligible.
* Organ allografts requiring immunosuppressive therapy.
* Serious uncontrolled intercurrent infections or other serious uncontrolled concomitant disease.
* Moderate or severe renal impairment [creatinine clearance equal to or below 50 ml/min (calculated according to Cockroft and Gault)], or serum creatinine > 1.5 x upper limit of normal (ULN).
* Any of the following laboratory values:

  * Absolute neutrophil count (ANC) < 1.5 x 109/L
  * Platelet count < 100 x 109/L
  * Total bilirubin > 1.5 x ULN
  * ALAT, ASAT > 2.5 x ULN
  * Alkaline phosphatase > 2.5 x ULN.
* Prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented dihydropyrimidine dehydrogenase (DPD) deficiency) or patients with known DPD deficiency.
* Hypersensitivity to platinum compounds or any of the components of the study medications.
* Received any investigational drug or agent/procedure, i.e. participation in another trial, within 4 weeks before randomization.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-09; Primary Completion 2020-08 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
3-year DFS | 3 years after surgery

SECONDARY OUTCOMES:
adverse events | From date of randomization until the end of the study, assessed up to 5 years
response rate | evaluate after the end of neoadjuvant chemotherapy ie within 1 weeks after the neoadjuvant therapy
R0 resection rate | after the pathological examination of resected speciments ie within 1 month after the operation
overall survival | 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yingwei Xue, Phd, MD, Study Director — Harbin Medical University
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China